CLINICAL TRIAL: NCT05868525
Title: Pilot, Non-masked, Randomized Clinical Trial for Evaluation of Stroke Rate in Patients With Blunt Cerebrovascular Injury (BCVI) Treated With Oral Acetylsalicylic Acid (ASA) 81 mg Versus ASA 325 mg (BASA).
Brief Title: Stroke Rate in Patients With Blunt Cerebrovascular Injury (BCVI) Treated With Oral Acetylsalicylic Acid (ASA) 81 mg Versus ASA 325 mg (BASA).
Acronym: BASA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5220429
Record Dates: First submitted 2023-05-01; First posted 2023-05-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Blunt Cerebrovascular Injury
Keywords: Blunt cerebrovascular injury; BCVI; Carotid artery; Vertebral Artery; Internal Carotid Artery
MeSH Terms: interventions — Aspirin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Daily Aspirin 81 mg (Active Comparator)
  Interventions: Drug: Aspirin 325Mg Tab, Aspirin 81Mg Tab
- Oral Daily Aspirin 325 mg (Active Comparator)
  Interventions: Drug: Aspirin 325Mg Tab, Aspirin 81Mg Tab

INTERVENTIONS:
Drug: Aspirin 325Mg Tab, Aspirin 81Mg Tab — Patients will be administrated daily oral Aspirin 81 mg or oral Aspirin 325 mg according to their assigned group after randomization.

SUMMARY:
The goal of this clinical trial is to compare difference between Aspirin 81 mg and Aspirin 325 mg in preventing strokes in patients with head and neck vessels injury.

The main questions it aims to answer are:

* If Aspirin 81 mg efficacy in prevention of stroke in patients with head and neck vessels injury is not lower than and Aspirin 325 mg.
* If rate of hemorrhagic complications in patients with head and neck vessels injury taking Aspirin 81 mg is not higher than patients that take Aspirin 325 mg.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* All patients with blunt cerebrovascular injury are diagnosed by computed tomography angiography (CTA) upon admission

Exclusion Criteria:

* Age <18
* Pregnant women
* No enteral route access for Aspirin administration
* Patients who are on Heparin drip or other full dose anticoagulation when BCVI diagnosed
* Patients who are on other Anti-Platelets aside from Aspirin when BCVI diagnosed
* Patients with BCVI grade 5 injury based on Biffl classification
* Presence of any contraindication or history of allergy to Aspirin
* Patient with the diagnosis of acute stroke at the time of BCVI diagnosis matching the injured vessel territory on imaging
* Patients with acute spinal trauma that needs surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with new stroke event (ischemic stroke or hemorrhagic stroke) | From randomization up to 3 months after discharge

SECONDARY OUTCOMES:
Number of patients that experienced any Aspirin-related adverse events | From randomization up to 3 months after discharge
  An allergic reaction or gastrointestinal bleeding
Rate of need for bleeding control operations/interventions in patients with solid organ injury | From randomization up to 30 day after randomization
Need for blood product transfusion | From randomization up to 30 day after randomization
Rate of any bleeding incidence | From randomization up to 30 day after randomization
  major or minor bleeds define according to the International Society of Thrombosis and Hemostasis (ISTH)
Number of patients that experienced any incidence of worsening brain hemorrhage | From randomization up to 30 day after randomization
Any change in the percentage (%) of luminal stenosis in injured vessels of the neck and head | From randomization up to 3 months after discharge
Change in severity of the neck and head vessels injury based on Biffl grading scale | From randomization up to 3 months after discharge
In-hospital mortality rate | From randomization up to 30 day after randomization
Out-patient mortality rate | From discharge up to 3 months after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brommeland T, Helseth E, Aarhus M, Moen KG, Dyrskog S, Bergholt B, Olivecrona Z, Jeppesen E. Best practice guidelines for blunt cerebrovascular injury (BCVI). Scand J Trauma Resusc Emerg Med. 2018 Oct 29;26(1):90. doi: 10.1186/s13049-018-0559-1. PMID 30373641
- [Background] Miller PR, Fabian TC, Croce MA, Cagiannos C, Williams JS, Vang M, Qaisi WG, Felker RE, Timmons SD. Prospective screening for blunt cerebrovascular injuries: analysis of diagnostic modalities and outcomes. Ann Surg. 2002 Sep;236(3):386-93; discussion 393-5. doi: 10.1097/01.SLA.0000027174.01008.A0. PMID 12192325
- [Background] Miller PR, Fabian TC, Bee TK, Timmons S, Chamsuddin A, Finkle R, Croce MA. Blunt cerebrovascular injuries: diagnosis and treatment. J Trauma. 2001 Aug;51(2):279-85; discussion 285-6. doi: 10.1097/00005373-200108000-00009. PMID 11493785
- [Background] Griffin RL, Falatko SR, Aslibekyan S, Strickland V, Harrigan MR. Aspirin for primary prevention of stroke in traumatic cerebrovascular injury: association with increased risk of transfusion. J Neurosurg. 2018 May 18;130(5):1520-1527. doi: 10.3171/2017.12.JNS172284. Print 2019 May 1. PMID 29775142
- [Background] Catapano JS, Israr S, Whiting AC, Hussain OM, Snyder LA, Albuquerque FC, Ducruet AF, Nakaji P, Lawton MT, Weinberg JA, Zabramski JM. Management of Extracranial Blunt Cerebrovascular Injuries: Experience with an Aspirin-Based Approach. World Neurosurg. 2020 Jan;133:e385-e390. doi: 10.1016/j.wneu.2019.09.013. Epub 2019 Sep 12. PMID 31521761
- [Background] Cothren CC, Biffl WL, Moore EE, Kashuk JL, Johnson JL. Treatment for blunt cerebrovascular injuries: equivalence of anticoagulation and antiplatelet agents. Arch Surg. 2009 Jul;144(7):685-90. doi: 10.1001/archsurg.2009.111. PMID 19620551
- [Background] Shahan CP, Magnotti LJ, McBeth PB, Weinberg JA, Croce MA, Fabian TC. Early antithrombotic therapy is safe and effective in patients with blunt cerebrovascular injury and solid organ injury or traumatic brain injury. J Trauma Acute Care Surg. 2016 Jul;81(1):173-7. doi: 10.1097/TA.0000000000001058. PMID 27027559
- [Background] McNutt MK, Kale AC, Kitagawa RS, Turkmani AH, Fields DW, Baraniuk S, Gill BS, Cotton BA, Moore LJ, Wade CE, Day A, Holcomb JB. Management of blunt cerebrovascular injury (BCVI) in the multisystem injury patient with contraindications to immediate anti-thrombotic therapy. Injury. 2018 Jan;49(1):67-74. doi: 10.1016/j.injury.2017.07.036. Epub 2017 Jul 31. PMID 28789779
- [Background] Callcut RA, Hanseman DJ, Solan PD, Kadon KS, Ingalls NK, Fortuna GR, Tsuei BJ, Robinson BR. Early treatment of blunt cerebrovascular injury with concomitant hemorrhagic neurologic injury is safe and effective. J Trauma Acute Care Surg. 2012 Feb;72(2):338-45; discussion 345-6. doi: 10.1097/TA.0b013e318243d978. PMID 22327975
- [Background] Biffl WL, Cothren CC, Moore EE, Kozar R, Cocanour C, Davis JW, McIntyre RC Jr, West MA, Moore FA. Western Trauma Association critical decisions in trauma: screening for and treatment of blunt cerebrovascular injuries. J Trauma. 2009 Dec;67(6):1150-3. doi: 10.1097/TA.0b013e3181c1c1d6. No abstract available. PMID 20009659
- [Background] Harrigan MR, Weinberg JA, Peaks YS, Taylor SM, Cava LP, Richman J, Walters BC. Management of blunt extracranial traumatic cerebrovascular injury: a multidisciplinary survey of current practice. World J Emerg Surg. 2011 Apr 8;6:11. doi: 10.1186/1749-7922-6-11. PMID 21477304
- [Background] Biffl WL, Moore EE, Ryu RK, Offner PJ, Novak Z, Coldwell DM, Franciose RJ, Burch JM. The unrecognized epidemic of blunt carotid arterial injuries: early diagnosis improves neurologic outcome. Ann Surg. 1998 Oct;228(4):462-70. doi: 10.1097/00000658-199810000-00003. PMID 9790336
- [Background] Malhotra A, Wu X, Seifert K, Tu L. Blunt Cerebrovascular Artery Injury and Stroke in Severely Injured Patients: An International Multicenter Analysis. World J Surg. 2018 Oct;42(10):3451. doi: 10.1007/s00268-018-4518-9. No abstract available. PMID 29383427
- [Background] Harrigan MR, Hadley MN, Dhall SS, Walters BC, Aarabi B, Gelb DE, Hurlbert RJ, Rozzelle CJ, Ryken TC, Theodore N. Management of vertebral artery injuries following non-penetrating cervical trauma. Neurosurgery. 2013 Mar;72 Suppl 2:234-43. doi: 10.1227/NEU.0b013e31827765f5. No abstract available. PMID 23417194
- [Background] DuBose J, Recinos G, Teixeira PG, Inaba K, Demetriades D. Endovascular stenting for the treatment of traumatic internal carotid injuries: expanding experience. J Trauma. 2008 Dec;65(6):1561-6. doi: 10.1097/TA.0b013e31817fd954. PMID 19077655